CLINICAL TRIAL: NCT05317676
Title: Effect of Palmitoylethanolamide on Reducing Opioid Consumption for Postoperative Pain and Inflammation Following Below Knee Fracture Fixation: A Pilot Study.
Brief Title: Effect of Palmitoylethanolamide on Reducing Opioid Consumption for Below Knee Fracture Fixation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor suspending temporarily.
Sponsor: University of California, Irvine (Other)
Collaborators: GE Nutrients Inc. (Gencor) (Unknown)
Responsible Party: Principal Investigator, Ariana M. Nelson, Associate Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-6007
Record Dates: First submitted 2022-02-22; First posted 2022-04-08 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Tibial Fractures; Fibula Fracture; Knee Fracture
Keywords: Palmitoylethanolamide; Open reduction and internal fixation (ORIF) Surgery; Postoperative Pain; Inflammation; Reduce Opioid Consumption
MeSH Terms: conditions — Tibial Fractures; Fibula Fractures; Knee Fractures; Pain, Postoperative; Inflammation | interventions — palmidrol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Palmitoylethanolamide (Active Comparator): 300 mg PEA twice a day for a total of 600 mg PEA daily 2-month supply upon discharge
  Interventions: Drug: Palmitoylethanolamide
- Placebo (Placebo Comparator): 1 placebo tablet twice a day for a total of 2 tablet placebo daily 2-month supply upon discharge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Palmitoylethanolamide — 2-month supply of PEA will be given upon discharge. 300mg will be taken twice a day in conjunction with discharge medications (opioid and NSAIDs).
  Other Names: PEA; GenCor
  Arms: Palmitoylethanolamide
Drug: Placebo — 2-month supply of placebo will be given upon discharge. Placebo will taken twice a day in conjunction with discharge medications (opioid and NSAIDs).
  Arms: Placebo

SUMMARY:
Palmitoylethanolamide (PEA), a non-psychoactive cannabis compound derived from peanuts, egg yolks, and soybeans, is an Endogenous FA Amide produced in the body as a biological response and a repair mechanism in chronic inflammation and chronic pain. In animal and clinical trials, PEA has also shown evidence of pain reduction, sleep improvement, and increased joint mobility and function with minimal side-effects. The study team intends to study whether the inclusion of PEA in conjunction with standard post-surgical medications can reduce pain and inflammation while decreasing the number of opioids needed.

DETAILED DESCRIPTION:
According to the National Center for Health Statistics, the United States sees approximately 492,000 tibial fractures per year. Of that population, there are greater than 70,000 hospitalizations, 800,000 office visits, and 500,000 hospital days attributed annually. This does not include the approximately 250,000 proximal femur fractures that occur in the US annually, which is expected to double by 2050. There are also over 5 million ankle injuries in the US per year at a rate of approximately 187 ankle fractures per 100,000 people. To repair these below knee fractures, patients with severe cases often have an open reduction and internal fixation (ORIF) surgery to stabilize and heal the broken bone.

On average, these patients are seen by physical therapy to determine their safety for going home and if they need any equipment like a walker or crutches. They are discharged with pain medications, such as analgesic opioids and stool softeners. These patients return to clinic in 2 weeks for follow up which involves an exam, suture removal, x-rays, and possibly weight bearing status update. They then return in 1 month for exam, x-rays, and weightbearing status. Finally they return at 3 months for exam, x-rays, and weightbearing status.

The study team intends to study whether the inclusion of PEA in conjunction with standard post-surgical medications can reduce pain and inflammation while decreasing the number of opioids needed

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Has an isolated below knee orthopaedic injury without any neurovascular injury involvement
* Has an isolated active orthopaedic injury
* Females of childbearing potential must have a negative urine and blood pregnancy test at Screening and a negative urine pregnancy test on Day 1 before study drug is administered. Females must abstain from sex or use a highly effective method of contraception during the period from Screening to administration of study drug and for 30 days after the last dose of study medication. Standard acceptable methods include abstinence or the use of a highly effective method of contraception, including; hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom with spermicide, vasectomy, intrauterine device.
* If females are of non-child bearing potential, they must be post-menopausal defined as: age > 55 with no menses within the past 12 months or history of hysterectomy, or history of bilateral oophorectomy, or bilateral tubal ligation.

Exclusion Criteria:

* Less than 18 years of age
* Pregnant or Breastfeeding
* Allergic to cannabis
* History of chronic opioid use
* History of substance abuse
* History of chronic use of cannabis products of any kind
* Has multiple active orthopaedic injuries
* Has neurovascular injury associated with your orthopaedic injury
* History of a syndrome that causes chronic pain (i.e. fibromuscular dysplasia, complex pain syndrome)
* History of peripheral neuropathy
* History of diagnosed psychiatric illness
* ASA score of greater than 3
* Clinically significant unstable medical condition, including but not limited to cardiovascular, neurologic, psychiatric, endocrine, hepatic, and renal disorders.
* Allergy to palmitoylethanolamide (PEA) or its derivatives such as soy or eggs
* AST/ALT ≥3x ULN and/or bilirubin ≥2x ULN at screening.
* Abnormal creatinine or renal function abnormalities.
* Have end stage organ failure (Cardiac, Renal, or Hepatic)
* Currently undergoing addiction/detoxification therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
3 month post-surgical Opioid use Questionnaire | 3 months
  Questionnaire (during call) asking patient for list of medications taken in last 2 days and cross referencing with opioid prescription in chart
3 month post-surgical NSAID use Questionnaire | 3 months
  Questionnaire (during call) asking patient for list of medications taken in last 2 days and cross referencing with NSAID prescription in chart

SECONDARY OUTCOMES:
Pain Scores | 3 months
  Pain scores using McGill Pain Questionnaire; minimum pain score: 0 (would not be seen in a person with true pain);maximum pain score: 78;The higher the pain score the greater the pain.
Pain Interference | 3 months
  Pain interference using PROMIS Pain Interference Survey; Each question usually has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 6-item form, the lowest possible raw score is 6; the highest possible raw score is 30.Locate the applicable score conversion table and use this table to translate the total raw score into a T-score for each participant. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10
Average Pain Scores | 3 months
  Pain scores using Brief Pain Inventory; 0-10 numerical rating scale used to measure three pain severity items: "worst" in the past month, "average," and "now," where 0=no pain and 10=pain as bad as you can imagine.
Functional Status | 3 months
  Functional status using PROMIS Physical Function Survey; The PF-10a is a 10-item questionnaire assessing current self-reported physical function. Raw scores range from 10 to 50 and can be translated into T-scores, with a mean of 50 and a standard deviation of 10, for comparison with the U.S. general population mean; for this study, all reported PF-10a scores are T-scores.
Post-Surgical Complications | 3 months
  Any complications following surgery
Medication Adverse Events | 3 months
  Any adverse events to study drug and post-surgical medications given at discharge
Average Pain Interference | 3 months
  Pain interference using Brief Pain Inventory; 0-10 numerical rating scale used to measure three pain severity items: "worst" in the past month, "average," and "now," where 0=no pain and 10=pain as bad as you can imagine.

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Nelson, MD, Principal Investigator — Associate Clinical Professor
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

REFERENCES:
- [Background] Artukoglu BB, Beyer C, Zuloff-Shani A, Brener E, Bloch MH. Efficacy of Palmitoylethanolamide for Pain: A Meta-Analysis. Pain Physician. 2017 Jul;20(5):353-362. PMID 28727699
- [Background] Grotenhermen F. Cannabinoids and the endocannabinoid system. Cannabinoids.2006;1:10-14.
- [Background] Martin-Sanchez E, Furukawa TA, Taylor J, Martin JL. Systematic review and meta-analysis of cannabis treatment for chronic pain. Pain Med. 2009 Nov;10(8):1353-68. doi: 10.1111/j.1526-4637.2009.00703.x. Epub 2009 Sep 1. PMID 19732371
- [Background] Cabral GA, Griffin-Thomas L. Emerging role of the cannabinoid receptor CB2 in immune regulation: therapeutic prospects for neuroinflammation. Expert Rev Mol Med. 2009 Jan 20;11:e3. doi: 10.1017/S1462399409000957. PMID 19152719
- [Background] Calignano A, La Rana G, Giuffrida A, Piomelli D. Control of pain initiation by endogenous cannabinoids. Nature. 1998 Jul 16;394(6690):277-81. doi: 10.1038/28393. PMID 9685157
- [Background] Calignano A, La Rana G, Piomelli D. Antinociceptive activity of the endogenous fatty acid amide, palmitylethanolamide. Eur J Pharmacol. 2001 May 11;419(2-3):191-8. doi: 10.1016/s0014-2999(01)00988-8. PMID 11426841
- [Background] Esposito E, Paterniti I, Mazzon E, Genovese T, Di Paola R, Galuppo M, Cuzzocrea S. Effects of palmitoylethanolamide on release of mast cell peptidases and neurotrophic factors after spinal cord injury. Brain Behav Immun. 2011 Aug;25(6):1099-112. doi: 10.1016/j.bbi.2011.02.006. Epub 2011 Feb 25. PMID 21354467
- [Background] Luongo L, Guida F, Boccella S, Bellini G, Gatta L, Rossi F, de Novellis V, Maione S. Palmitoylethanolamide reduces formalin-induced neuropathic-like behaviour through spinal glial/microglial phenotypical changes in mice. CNS Neurol Disord Drug Targets. 2013 Feb 1;12(1):45-54. doi: 10.2174/1871527311312010009. PMID 23394524
- [Background] Scuderi C, Steardo L. Neuroglial roots of neurodegenerative diseases: therapeutic potential of palmitoylethanolamide in models of Alzheimer's disease. CNS Neurol Disord Drug Targets. 2013 Feb 1;12(1):62-9. doi: 10.2174/1871527311312010011. PMID 23394526
- [Background] Nau R, Djukic M, Spreer A, Ribes S, Eiffert H. Bacterial meningitis: an update of new treatment options. Expert Rev Anti Infect Ther. 2015;13(11):1401-23. doi: 10.1586/14787210.2015.1077700. Epub 2015 Aug 18. PMID 26293166
- [Background] Gabrielsson L, Mattsson S, Fowler CJ. Palmitoylethanolamide for the treatment of pain: pharmacokinetics, safety and efficacy. Br J Clin Pharmacol. 2016 Oct;82(4):932-42. doi: 10.1111/bcp.13020. Epub 2016 Jun 29. PMID 27220803
- [Background] COBURN AF, GRAHAM CE, HANINGER J. The effect of egg yolk in diets on anaphylactic arthritis (passive Arthus phenomenon) in the guinea pig. J Exp Med. 1954 Nov 1;100(5):425-35. doi: 10.1084/jem.100.5.425. PMID 13211905
- [Background] Hesselink JM. Evolution in pharmacologic thinking around the natural analgesic palmitoylethanolamide: from nonspecific resistance to PPAR-alpha agonist and effective nutraceutical. J Pain Res. 2013 Aug 8;6:625-34. doi: 10.2147/JPR.S48653. eCollection 2013. PMID 23964161